CLINICAL TRIAL: NCT00018603
Title: Guanfacine for the Treatment of PTSD
Brief Title: Guanfacine for the Treatment of Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS-047-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Guanfacine

INTERVENTIONS:
Drug: guanfacine

SUMMARY:
This is a double-blind, placebo-controlled, randomized study lasting 8 weeks. Purpose of the study is two-fold: first, to use a pharmacological agent to treat symptoms of PTSD, and second, to explore neurobiological mechanisms of action of guanfacine.

DETAILED DESCRIPTION:
Subject population is comprised of 100 persons with PTSD. 50 patients will receive guanfacine and 50 patients will receive a placebo. Guanfacine is prescribed at 1 mg/day and may be increased to 2 mg/day. Samples of plasma MHPG will be collected weekly. Clinical ratings of PTSD anxiety and depression, as well as vital signs, will be assessed weekly. Repeated measures analysis of variance will assess significance of main effect of drug, time, and drug by time.

ELIGIBILITY:
* Males and females, age 18-65
* Diagnosis of PTSD from combat or civilian trauma
* No major medical problems such as diabetes, cardiovascular disease
* Taking no psychiatric medication, or taking only one SSRI antidepressant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States